CLINICAL TRIAL: NCT01015586
Title: A Double-Blind, Placebo-Controlled Trial of Lamotrigine In Individuals With Bipolar Disorder and Comorbid Alcohol Dependence
Brief Title: Treatment of Alcohol Dependence and Comorbid Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HR#19550; K23AA017666 (NIH)
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Results first posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Alcohol Dependence; Bipolar Disorder; Depression; Mania; Psychosis
Keywords: Alcohol; Bipolar Disorder; Manic depression; Addiction; Alcoholism; Cognitive impairment; Executive function; Anxiety; Depression; Mania; Affective disorder; Psychosis; Carbohydrate deficient transferrin; Gammaglutamyltransferase; California Verbal Learning Test; Montgomery Asberg Depression Rating Scale; Young Mania Rating Scale; Timeline Follow Back
MeSH Terms: conditions — Alcoholism; Bipolar Disorder; Depression; Mania; Psychotic Disorders; Behavior, Addictive; Cognitive Dysfunction; Anxiety Disorders; Mood Disorders | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lamotrigine (Experimental): Add-on lamotrigine plus pre-existing mood stabilizing medication regimen. Active fixed-dose drug titration from 25-200 mg/day over first six weeks, 200 mg/day fixed-dose maintenance for second six weeks
  Interventions: Drug: Lamotrigine
- Placebo (Placebo Comparator): Add-on placebo plus pre-existing mood stabilization regimen for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lamotrigine — Six week titration from 25 mg/day to 200 mg/day, then 200 mg/day maintenance for additional six weeks
  Arms: Lamotrigine
Drug: Placebo — Placebo once daily for 12 weeks
  Arms: Placebo

SUMMARY:
The study will determine if individuals with co-occurring bipolar disorder and alcohol dependence report reduced alcohol consumption, improvement in mood symptoms, and cognitive performance if treated with lamotrigine plus their usual mood stabilizing medications relative to subjects treated with placebo plus usual mood stabilizing medications over a 16 week period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Meet DSM-IV-TR criteria for current alcohol dependence with active alcohol use in the past 30 days
* Meet DSM-IV-TR criteria for bipolar I or bipolar II disorder
* Have average alcohol consumption of at least 35 drinks/week for men, 28 drinks/week for women in the last 4 weeks of active drinking prior to enrollment.
* Able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of the assessment instruments.
* Must consent to random assignment and be willing to commit to medication treatment and follow-up assessments.
* Currently under the care of a psychiatrist.
* Must consent to sign a release of information allowing investigators to communicate with his/her psychiatrist to verify treatment history and facilitate care should treatment-emergent psychiatric symptoms develop during the trial.
* Currently taking a therapeutic dosage of one or more mood stabilizing medications as defined by one or more of the following:

  * Lithium level of 0.6 - 1.2 mEq/L
  * Prescribed daily use of first generation antipsychotic agents including chlorpromazine, fluphenazine, or haloperidol or their injectible depot (decanoate) equivalents at a dose adequate to maintain clinical stability as documented by the subject's outpatient psychiatric provider c) Prescribed daily use of second generation antipsychotic agents including olanzapine, risperidone, paliperidone, quetiapine, aripiprazole, or ziprasidone or their injectible depot equivalent at a dose adequate to maintain clinical stability as documented by the subject's outpatient psychiatric provider
* Stable psychiatric symptoms as defined by no changes to psychotropic drug regimen for 30 days
* Must agree to identify collateral individuals for contact to facilitate follow-up appointments

Exclusion Criteria:

* A primary psychiatric diagnosis other than bipolar disorder
* Any uncontrolled neurologic condition (e.g. epilepsy) that could confound the results of the study
* Any history of Stevens-Johnson syndrome or other severe rash requiring hospitalization
* Any history of head injury with loss of consciousness greater than 30 minutes
* Any history of learning disability, alcoholic dementia, or electroconvulsive therapy in the past 3 months
* Any uncontrolled medical condition that may adversely affect the conduct of the trial or jeopardize the safety of the subject
* Plasma levels of liver transaminases (AST, ALT) greater than 3 times the normal range
* Concomitant use of valproic acid
* Concomitant use of carbamazepine, oxcarbazepine, phenytoin, primidone, or phenobarbital
* Concomitant use of disulfiram, naltrexone, acamprosate, or topiramate
* Concomitant use of benzodiazepines or any other medications not allowed per the protocol
* Women of childbearing potential who are pregnant, lactating, or refuse adequate forms of contraception
* Current suicidal or homicidal risk
* Baseline scores of more than 35 on the Montgomery-Asberg Depression Rating Scale or more than 16 on the Young Mania Rating Scale

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-02; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan K Tolliver, MD, PhD, Principal Investigator — Medical University of South Carolina; Kathleen T Brady, M.D., Ph.D., Study Director — Medical University of South Carolina
Locations (1):
- Clinical Neuroscience Division, Department of Psychiatry and Behavioral Sciences, Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lamotrigine | Placebo
Started | 21 | 22
Completed | 14 | 11
Not Completed | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lamotrigine | Placebo | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.48 (11.46) | 44.14 (10.13) | 44.30 (10.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 15 | 15 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 16 | 20 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 22 | 43

OUTCOME MEASURES:

1. Primary Outcome: Percent Days Abstinent From Alcohol
Description: Percentage of days in trial without consumption of alcoholic beverages per participant self-report; minimum = 0, maximum = 100; higher numbers indicate better outcome. Percent days abstinent was calculated as: (number of days abstinent per self-report / total number of days in trial)*100.
Time Frame: 12 weeks
Population: Analysis is of modified intention to treat (ITT) sample comprised of all randomized subjects who returned for at least one study visit after randomization.
Measure: Mean (Standard Deviation); unit: Percentage of days abstinent
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 20 | 17
Percentage of days abstinent | 78.7 (30.0) | 80.1 (28.4)

2. Secondary Outcome: Percent Heavy Drinking Days
Description: Percentage of days in trial that were heavy drinking days (5 or more drinks/day for men, 4 or more drinks/day for women); minimum = 0, maximum = 100; lower numbers indicate better outcome. Percent heavy drinking days was calculated as: (number of days of heavy drinking per self-report / total number of days in trial)*100.
Time Frame: 12 weeks
Population: Analysis is of modified intention to treat (mITT) sample comprised of all randomized subjects who returned for at least one study visit after randomization (total mITT sample n=37).
Measure: Mean (Standard Deviation); unit: Percentage of heavy drinking days
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 20 | 17
Percentage of heavy drinking days | 8.1 (12.8) | 11.6 (21.1)

3. Secondary Outcome: Biomarkers of Alcohol Use: Carbohydrate-deficient Transferrin (CDT)
Description: Serum levels of biomarkers of alcohol use: carbohydrate-deficient transferrin (CDT) at study endpoint in study completers
Time Frame: 12 weeks after randomization
Population: The sample analyzed is limited to study completers (total n=25) due to this measure being obtained at study endpoint.
Measure: Mean (Standard Deviation); unit: "percent CDT"
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 13 | 12
"percent CDT" | 1.41 (.48) | 1.26 (.18)

4. Secondary Outcome: Biomarkers of Alcohol Use: Gamma-glutamyltransferase (GGT)
Description: Serum levels of biomarkers of alcohol use: Gamma-glutamyltransferase (GGT) at study endpoint in study completers
Time Frame: 12 weeks after randomization
Population: Sample in this analysis is limited to study completers only (total n=25) because this measure was obtained at study endpoint.
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 13 | 12
Units per liter (U/L) | 62.5 (139.4) | 22.9 (10.7)

5. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Score
Description: Scores on the Montgomery-Asberg Depression Rating Scale (MADRS) at baseline (all randomized subjects) and at study endpoint (study completers). Scores represent total summed score of ten (10) subscale items; minimum = 0, maximum = 60, higher scores indicate worse outcomes.
Time Frame: Baseline and 12 weeks
Population: All randomized subjects (total n=43) included in analysis at baseline. Study completers only (total n=25) included in analysis at study endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 21 | 22
units on a scale
  Baseline MADRS score | 9.86 (5.34) | 12.05 (6.21)
  MADRS score at study endpoint: number analyzed (Participants) | 13 | 12
  MADRS score at study endpoint | 6.93 (5.36) | 9.18 (5.67)

6. Secondary Outcome: Young Mania Rating Scale (YMRS) Scores
Description: Mania/hypomania symptoms at study endpoint as assessed by the Young Mania Rating Scale (YMRS) at baseline (all randomized subjects) and at study endpoint (study completers). Scores represent total summed score of eleven (11) subscale items; minimum = 0, maximum = 60, higher scores indicate worse outcomes.
Time Frame: Baseline and 12 weeks
Population: Baseline YMRS scores include all randomized subjects (total n=43). Study endpoint YMRS scores include study completers only (total n=25).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 21 | 22
score on a scale
  Baseline YMRS scores | 7.30 (4.50) | 9.25 (5.58)
  Endpoint YMRS scores: number analyzed (Participants) | 13 | 12
  Endpoint YMRS scores | 5.50 (2.65) | 7.40 (4.03)

7. Secondary Outcome: Neurocognitive Performance (California Verbal Learning Test)
Description: Adjusted scale scores (T scores) on the California Verbal Learning Test (CVLT) of verbal working memory at study endpoint. CVLT Trials 1-5 Free Recall Total measures the sum of all word list items correctly recalled on learning trials 1 through 5. This raw score is converted to a T-score (mean = 50; SD=10) with higher scores indicating better performance.
Time Frame: Study endpoint 12 weeks after randomization
Population: Sample analyzed includes study completers only (total n=25) as this measure was obtained at study endpoint.
Measure: Mean (Standard Deviation); unit: T scores
Arm/Group | Lamotrigine | Placebo
Number analyzed (Participants) | 13 | 12
T scores | 58.9 (14.6) | 52.1 (12.5)

ADVERSE EVENTS:
Time Frame: 18 weeks (two-week baseline assessment phase, 12 week active medication phase, 4 week safety phase after medication discontinuation)
Arm/Group | Lamotrigine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/21 | 1/22
Other Adverse Events (participants affected / at risk) | 9/21 | 9/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lamotrigine (N=21) | Placebo (N=22)
Hospitalization (Psychiatric disorders) | 1 (1) | 1 (1) — Active suicidal ideation with plan to overdose on medications
Hospitalization (medical) after assault (Surgical and medical procedures) | 0 (0) | 1 (1) — Neurosurgical evacuation of epidural hematoma, intensive care required after serious assault
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lamotrigine (N=21) | Placebo (N=22)
Headache (General disorders) | 3 (3) | 1 (1)
Erythema / skin discoloration (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Papular skin eruption (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Flu-like symptoms (General disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Relatively small sample size, suboptimal retention rate (58% of all randomized subjects)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No